CLINICAL TRIAL: NCT01664169
Title: Validation of Circulating Biomarkers Using the Immunological Multiparameter Chip Technology (IMPACT) on Plasma Specimens Collected on CALGB 80303
Brief Title: Biomarkers in Plasma Specimens From Patients Treated on Study CALGB-80303
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: A151201; CDR0000738204 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-01994 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; stage IIB pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The following markers are analyzed in EDTA plasma samples using the IMPACT a Roche proprietary multiplex ELISA platform: VEGF-A, VEGF-C, VEGF-R1, VEGF-R2, E-selectin, VEGF-R3, IL-8, bFGF, PDGF-C, ICAM-1, and PlGF.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group: The samples required for this study are stored in the CALGB Pathology Coordinating Office at The Ohio State University from patients enrolled on protocol CALGB-80303. No additional samples are required from patients.
  The following markers are analyzed in EDTA plasma samples using the IMPACT a Roche proprietary multiplex ELISA platform: VEGF-A, VEGF-C, VEGF-R1, VEGF-R2, E-selectin, VEGF-R3, IL-8, bFGF, PDGF-C, ICAM-1, and PlGF.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying plasma samples from patients with pancreatic cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in samples from patients with pancreatic cancer treated on study CALGB-80303.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether the observed predictive value of plasma VEGF-A and VEGF-R2 for overall survival (OS) in study BO17706 can be replicated in study CALGB-80303 using the same Immunological Multiparameter Chip Technology (IMPACT) assay.
* To determine whether the observed predictive value of plasma VEGF-A and VEGF-R2 for progression-free survival (PFS), and other circulating biomarkers in study BO17706, can be replicated in study CALGB-80303 using the same IMPACT assay.
* To explore the relationship between efficacy and other biomarkers measured in the plasma samples.

OUTLINE: The samples required for this study are stored in the CALGB Pathology Coordinating Office at The Ohio State University from patients enrolled on protocol CALGB-80303. No additional samples are required from patients.

The following markers are analyzed in EDTA plasma samples using the Immunological MultiParameter Chip Technology (IMPACT) a Roche proprietary multiplex enzyme-linked immunosorbent assay (ELISA) platform: VEGF-A, VEGF-C, VEGF-R1, VEGF-R2, E-selectin, VEGF-R3, IL-8, bFGF, PDGF-C, ICAM-1, and PlGF.

ELIGIBILITY:
Patients must have been registered to CALGB-80303

* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* Locally advanced or metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pancreatic cancer and previously enrolled on CALGB-80303.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 month
Progression free survival | 1 month
Number and percentage of responder | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Pang, PhD, Principal Investigator — CALGB Statistical Office at Duke University Medical Center